CLINICAL TRIAL: NCT00121745
Title: Phase I Evaluation of Safety of Intravenous Infusion of a Pathotropic Vector Bearing a Cytocidal Cyclin G1 Construct (Rexin-G) as Intervention for Locally Advanced and Metastatic Pancreatic Cancer Refractory to Standard Chemotherapy
Brief Title: Evaluation of Safety of Rexin-G Gene Transfer for Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Epeius Biotechnologies (Industry)
Responsible Party: Erlinda M. Gordon, M.D., Epeius Biotechnologies Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC044C
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Pancreatic Cancer
Keywords: gene transfer; cell cycle control; cancer gene therapy; pathotropic targeting; tumor targeted retroviral vector
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Genetic: Rexin-G Dose 1
- 2 (Experimental)
  Interventions: Genetic: Rexin-G Dose 2
- 3 (Experimental)
  Interventions: Genetic: Rexin-G Dose 3
- 4 (Experimental)
  Interventions: Genetic: Rexin-G Dose 4

INTERVENTIONS:
Genetic: Rexin-G Dose 1 — Dose Level # Patients Treatment Days Vector Dose/Day Max.Volume/Dose I 3- 6 Days 1-7, 15-21 7.5 x 10e9 cfu 500 ml
  Arms: 1
Genetic: Rexin-G Dose 2 — Dose Level # Patients Treatment Days Vector Dose/Day Max.Volume/Dose II 3- 6 Days 1-7, 15-21 1.1 x 10e10 cfu 500 ml
  Arms: 2
Genetic: Rexin-G Dose 3 — Dose Level # Patients Treatment Days Vector Dose/Day Max.Volume/Dose
  III 3- 6 5 days/wk x 4 wks 3.0 x 10e10 cfu 500 ml
  Arms: 3
Genetic: Rexin-G Dose 4 — Dose Level # Patients Treatment Days Vector Dose/Day Max.Volume/Dose
  IV 3- 6 5 days/wk x 4 wks 8.0 x 10e10 cfu 500 ml
  Arms: 4

SUMMARY:
This is a dose-seeking study that will test the safety of increasing doses of Rexin-G, given intravenously, in patients with advanced or metastatic pancreatic cancer who have failed standard chemotherapy. Rexin-G is a tumor-targeted gene therapy vector that contains a "killer" gene that blocks the action of the human cyclin G1 gene. Cyclin G1 is a cell cycle control element that plays an important role in cancer growth. When injected into a vein, the Rexin-GTM vector seeks out and accumulates in cancerous tumors, therefore, increasing the concentration of the drug in the cancerous tumors and not in normal neighbouring organs.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer death in the United States. Every year, about 30,000 new patients are diagnosed with pancreatic cancer, and most will die within the year. The few patients that live beyond one year are those who have operable tumors whose cancer has not spread beyond the pancreas. There is no effective treatment for pancreatic cancer that impacts survival beyond a few more months. Therefore, innovative treatments are urgently needed. A number of experimental therapies are currently under investigation, and gene therapy is a viable therapeutic option.

A gene called cyclin G1 has been shown to play a very important part in cancer growth. In animal experiments, when this cyclin G1 gene is blocked, the cancer cells grow much slower or even die. This study will test the drug, Rexin-G, which contains a gene that works by getting rid of the cyclin G1 gene. The new gene will get into the tumor cells using a "vehicle" to carry it into the cells. The "vehicle" that will be used is a virus that has been changed so that it is not likely to cause disease. This "vehicle" is called a vector. When injected into a vein, the Rexin-G vector is designed to seek out and accumulate in cancerous tumors, therefore, increasing the concentration of the drug in the area of the cancer and not in normal neighbouring organs. When the killer gene gets into the cancer cell, it becomes part of the cell's genes and tells the cancer cell to begin using the new gene instead of the cyclin G1 gene. It is hoped that the Rexin-G will arrest the growth of the cancer or eradicate the tumor.

The goals of the study are to determine how much Rexin-G can be given to a patient, to assess how long Rexin-G stays in the body when injected into a vein, and if the drug would cause antibodies to form, transfer the gene to normal tissues or pass on the gene to another person or the person's offspring. The final goal is to determine if the Rexin-G vector can shrink the tumor by comparing the size of the tumor nodules measured by CT scan or MRI before and after the Rexin-G treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Locally advanced or metastatic pancreatic cancer.
* Histologic or cytologic confirmation at diagnosis or recurrence of pancreatic cancer
* Measurable disease (RECIST) criteria. Tumor lesions that are situated in a previously irradiated area are not considered measurable, except if there is radiologically confirmed progression of disease within the radiation fields after radiation was completed.
* Failed gemcitabine chemotherapy as indicated by disease progression ≤ 6 months from last gemcitabine treatment
* Two or less than 2 chemotherapy regimens for recurrent/progressive disease.
* Adequate hepatic function based on laboratory values obtained less than 7 days prior to registration:

  * Total bilirubin <2.0 mg/dL;
  * AST < 2 x ULN;
  * AST < 2 x ULN;
  * Hgb > 9.0 gm/dL;
  * PT < ULN;
  * PTT <ULN;
  * Albumin > 3.0 gm/dL;
  * Alkaline phosphatase < 3 x ULN;
  * Absolute granulocyte count > 1000/uL;
  * Platelet count > 100,000/uL;
  * Serum creatinine < 1.2 mg/dL for females; < 1.4 mg/dL for males.
* ECOG performance status (PS) 0 or 1.
* Ability to provide informed consent.
* Life expectancy 12 weeks or greater.
* Male participants should be willing to provide semen samples at required intervals. Inability of the patient to provide all semen samples does not make the patient ineligible. (EXCEPTION: If the patient has been vasectomized. To be noted in the study file).
* Fertile patients agree to use barrier contraception (condoms plus spermicidal jelly) during the vector infusion period and for six weeks after infusion.
* Accessibility of peripheral or central IV line which is adequate for infusions of investigational agent.

Exclusion Criteria:

* Prior malignancy. (EXCEPTION: Patients who are disease free ≥ 5 years and/or patients with non-melanoma skin cancer, Stage I breast cancer, CIS of cervix)
* Any of the following:

  * Pregnant women;
  * Nursing women;
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.). This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.
* Patients who are HIV+, HBV+ or HCV+.
* Clinically significant ascites causing symptoms or requiring therapeutic paracentesis.
* Medical, psychiatric, or social conditions that would compromise successful adherence to this protocol.
* Concomitant use of other chemotherapeutic, viral or immunotherapeutic agents is not allowed during the 6-week study period.
* ≤ 4 weeks from radiation therapy of their pancreatic primary or ≤ 2 weeks from palliative radiation therapy to metastatic sites.
* ≤ 4 weeks from prior chemotherapy.
* History of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicity and maximum tolerated dose of Rexin-G administered as intravenous infusions; To evaluate pharmacokinetics of Rexin-G | 22 months

SECONDARY OUTCOMES:
To assess anti-tumor activity of intravenously administered Rexin-G and obtain preliminary data on biochemical markers of tumor response | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, M.D., Principal Investigator — Mayo Clinic - Rochester, Minnesota
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States